CLINICAL TRIAL: NCT03183154
Title: Mathematical Modeling of the HIV Transmission Risk During the First 24 Weeks After Initiation of Antiretroviral Therapy in naïve HIV-infected MSM: Comparison of INSTI-based Regimens vs. nnRTI and PI Based Regimens.
Brief Title: Mathematical Modeling of the HIV Transmission Risk After Initiation of Antiretroviral Therapy in naïve HIV-infected
Acronym: MIAMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: University of California, Los Angeles (Other); J Parrondo Health (Unknown); Fundación para la Investigación Biomédica del Hospital Gregorio Maranon (Other)
Responsible Party: Sponsor
Other Study IDs: FIBHGM-EONC001-2016
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The objective of this study is to explore the impact of initiation of ART with different regimens in naïve MSM (in the setting of acute and chronic HIV-infection) on the probability of transmission of HIV by mathematical modeling.

DETAILED DESCRIPTION:
The HIV epidemic among men who have sex with men (MSM) continues to expand in low, middle, and high-income countries. The disproportionate HIV disease burden in MSM is explained largely by the high per act and per-partner transmission probability of HIV transmission in receptive anal sex . Current strategies are inadequate to control HIV spread among MSM; much more vigorous prevention efforts are required, including the early initiation of antiretroviral therapy (ART) that has been shown to reduce the rates of sexual transmission of HIV-1 and the adaptation and expanded use of pre-exposure prophylaxis (PrEP) to prevent the acquisition of HIV-1 infection .

Initiation of ART with regimens based on integrase strand transfer inhibitors (INSTI) is associated with a faster decline in HIV-RNA load than what is observed with regimens based on non-nucleoside transcriptase inhibitors (nnRTI), and protease inhibitors (PI). The clinical impact of this finding is unknown although clinical anecdotes suggest that it may it may cause a rapid decline in HIV RNA in women presenting with HIV in late pregnancy.

The objective of this study is to explore the impact of initiation of ART with different regimens in naïve MSM (in the setting of acute and chronic HIV-infection) on the probability of transmission of HIV by mathematical modeling.

ELIGIBILITY:
Inclusion Criteria:

* naïve HIV-infected MSM

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — men who have sex with men (MSM)
Study Population: naïve HIV-infected MSM
Sampling Method: Non-Probability Sample
Enrollment: 1831 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
To estimate the probability of HIV transmission during the first 24 weeks after initiation of cART in naïve HIV-infected MSM (in the setting of acute and chronic HIV-infection), with regimens based on nnRTI, INSTI, and PI | 24 weeks after initiation of cART
  1. To estimate the probability of HIV transmission during the first 24 weeks after initiation of cART in naïve HIV-infected MSM (in the setting of acute and chronic HIV-infection), with regimens based on nnRTI, INSTI, and PI

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berenguer J, Parrondo J, Landovitz RJ. Mathematical modeling of HIV-1 transmission risk from condomless anal intercourse in HIV-infected MSM by the type of initial ART. PLoS One. 2019 Jul 19;14(7):e0219802. doi: 10.1371/journal.pone.0219802. eCollection 2019. PMID 31323075